CLINICAL TRIAL: NCT05282251
Title: Pain Managment After VATS to Reduce Postoperative Pain and Improve Pulmonary Function
Brief Title: Intrapleural Nebulization of Bupivacain to Reduce Postoperative Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Essam El-den Moubark Mohammed Hussein, Resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pain managment after VATS
Record Dates: First submitted 2021-10-10; First posted 2022-03-16 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases | interventions — Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrapleural bupivacine nebulization (Experimental): Intrapleural nebulization of bupivacine (10 ml of bupivacaine 0.5%) + Intravenous normal saline as a placebo
  Interventions: Drug: Intrapleural bupivacine nebulization
- Intravenous paracetamol and ketorolac (Active Comparator): Intravenous analgesia: paracetamol (one gram) and Ketorolac (30 mg) + Intrapleural normal saline (10 ml) as a placebo
  Interventions: Drug: Intravenous paracetamol and ketorolac

INTERVENTIONS:
Drug: Intrapleural bupivacine nebulization — Intrapleural nebulization of bupivacine (10 ml of bupivacaine 0.5%) + Intravenous normal saline as a placebo
  Arms: Intrapleural bupivacine nebulization
Drug: Intravenous paracetamol and ketorolac — Intravenous analgesia: paracetamol (one gram) and Ketorolac (30 mg) + Intrapleural normal saline (10 ml) as a placebo
  Arms: Intravenous paracetamol and ketorolac

SUMMARY:
Thoracic surgery is now common and as other surgeries evolution of minimally invasive techniques is employed. Video-assisted thoracic surgery (VATS) produces little scar but may produce severe pain that may affect the pulmonary function. Many procedure was developed like intercostal nerve block which require injections at multiple levels, Insertion of local anaesthetic (LA) in the surgical drain but that was dangerous due to the large amount of LA and not sufficient to completely eliminate pain. Bupvicaine nebulization, through surgical port which won't make any other wound, thought to be sufficient because Nebulization will enable us better distribution and less amounts of LA. Bupvicaine is local anaesthetic amide group that works by blocking sodium channels thus preventing progression of action potential.

ELIGIBILITY:
Inclusion Criteria:

* Patients that reach American socity of anesthesiologist class 1-3
* Scheduled for VATS surgery under general anesthesia.

Exclusion Criteria:

* ● Allergy to local anesthetics

  * Patient with pleural inflammation due to recent pneumonia
  * Patients who are unable or unwilling to perform spirometer test
  * Renal dysfunction: (Elevated creatinine > 2 mg\dl)
  * Hepatic dysfunction: (Elevated hepatic enzymes three times above normal value)
  * History of addiction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Time to first rescue analgesia | The first 24 hours postoperatively

SECONDARY OUTCOMES:
Total opioid consumption | The first 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Assuit, Egypt